CLINICAL TRIAL: NCT01019499
Title: The Effect of Berry Consumption on Indicators of Cardiovascular Disease Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Finnish Institute for Health and Welfare (Other Government)
Collaborators: Agrifood Research Finland (Unknown); The Finnish Funding Agency for Technology and Innovation (TEKES) (Other Government); Academy of Finland (Other); University of Oslo (Other)
Responsible Party: Iris Erlund, Senior researcher, National Institute for Health and Welfare
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: NPHIKTL
Record Dates: First submitted 2009-11-24; First posted 2009-11-25 (Estimated); Last update posted 2010-06-22 (Estimated); Status verified 2010-06

CONDITIONS: Blood Pressure; Platelet Function; Inflammation
Keywords: human; intervention; blood pressure; cardiovascular risk factors; polyphenols; bioavailability
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- berry products (Active Comparator): Berry products
  Interventions: Other: berry products
- control products (Placebo Comparator): Control products
  Interventions: Other: control products

INTERVENTIONS:
Other: berry products — effects of berry consumption on cardiovascular indicators
  two portions daily
  Arms: berry products
Other: control products — two portions daily
  Arms: control products

SUMMARY:
The purpose of this study is to investigate the effects of berry consumption on indicators of cardiovascular disease risk (blood pressure, cardiovascular biomarkers, nutrigenomics).

DETAILED DESCRIPTION:
The study has a randomized crossover design. It consists of two 8-wk dietary treatments, with no washout period between periods. The participants are blinded to treatments. The subjects are randomly assigned to either a berry diet or a control diet which they follow for 8 weeks. After that they are crossed over to the other diet for another 8 weeks. The main visits to the study site are at baseline and after 8 and 16 weeks (for blood pressure measurement/ cardiovascular measurements and sample collection). The additional visits are at 4 and 12 wk; these visits are for compliance checks, meeting the study nurse and receiving the study products. The subjects are asked to maintain their normal dietary and lifestyle habits, as well as to keep alcohol intake and physical activity constant during the study.

ELIGIBILITY:
Inclusion Criteria:

* mild hypertension (systolic blood pressure 130-159 mmHg, diastolic blood pressure 85-99 mmHg)

Exclusion Criteria:

* smoking
* regular use of medications (except hormone replacement therapy) or dietary supplements
* intestinal disorders
* obesity (BMI> 35 kg/m2)
* vegetarianism
* pregnancy

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2009-02; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Blood pressure | 0, 8 and 16 weeks

SECONDARY OUTCOMES:
PFA-100 measurement | 0, 8 and 16 weeks
biomarkers of cardiovascular disease risk | 0, 8 and 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Antti Jula, DR., Study Director — Finnish Institute for Health and Welfare
Locations (2):
- Finland (2):
  - National Institute for Health and Welfare, Helsinki, Helsinki
  - National Institute for Health and Welfare, Turku, Turku